CLINICAL TRIAL: NCT03162094
Title: A Phase I/II, Double-blind, Placebo-controlled Study Assessing the Safety and Efficacy of AVX-012 Ophthalmic Solution in Subjects With Mild-to-moderate Dry Eye Syndrome
Brief Title: Assessing the Safety and Efficacy of AVX-012 in Subjects With Mild-to-moderate Dry Eye Syndrome
Acronym: AVX012CT001
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avizorex Pharma, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVX012 CT001; 2016-001022-34 (EudraCT Number)
Record Dates: First submitted 2017-04-05; First posted 2017-05-22 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Phase I: patient will be included on 3 arms of treatment ( Placebo, Low dose or High dose AVX-012) TID
  Phase II: Patient will be included on 4 arms of treatment (Placebo/Dose) BID/TID
Who Masked: Participant, Care Provider, Investigator
Masking Description: phase I/II, double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AVX-012 Opthalmic Solution Low dose (Experimental): Phase I: AVX-012 ophthalmic solution Low dose administration three times per day (TID) for 7 days
  Phase II: If the low dose of AVX012 is selected on phase I, AVX-012 ophthalmic solution Low dose administration three times per day (TID) and two times per day (BID) for 28 days
  Interventions: Drug: AVX012 Ophthalmic Solution Low dose
- AVX-012 Opthalmic Solution High dose (Experimental): Phase I: AVX-012 ophthalmic solution High dose administration three times per day (TID) for 7 days
  Phase II: If the high dose of AVX012 is selected on phase I, AVX-012 ophthalmic solution High dose administration three times per day (TID) and two times per day (BID) for 28 days
  Interventions: Drug: AVX012 Ophthalmic Solution High dose
- Placebo (Vehicle) Opthalmic Solution (Placebo Comparator): Phase I: Placebo ophthalmic solution administration three times per day (TID) for 7 days
  Phase II: Placebo ophthalmic solution administration three times per day (TID) and two times per day (BID) for 28 days
  Interventions: Drug: Placebo (vehicle)

INTERVENTIONS:
Drug: AVX012 Ophthalmic Solution Low dose — Ocular topical administration of AVX Ophthalmic Solution Low dose
  Arms: AVX-012 Opthalmic Solution Low dose
Drug: AVX012 Ophthalmic Solution High dose — Ocular topical administration of AVX Ophthalmic Solution High dose
  Arms: AVX-012 Opthalmic Solution High dose
Drug: Placebo (vehicle) — Ocular topical administration of placebo (vehicle Ophthalmic Solution)
  Arms: Placebo (Vehicle) Opthalmic Solution

SUMMARY:
This is a first-in-human phase I/II randomized, double-blind, placebo (vehicle)-controlled, multicenter study to assess the Safety and Efficacy of AVX-012 Ophthalmic Solution in subjects with Mild-to-Moderate Dry Eye Syndrome.

The study consists of two parts (part A and part B):

DETAILED DESCRIPTION:
The study part A will be an early safety assessment of AVX-012 ophthalmic solution (Low dose and High dose AVX-012) administered three times per day (TID) when compared with the vehicle (placebo). Approximately 24 patients will be randomized 1:1:1 to study groups (Low dose AVX-012, High dose AVX-012, or placebo [vehicle]).

An independent safety committee will be in charge of assessing the safety of study treatments to proceed to part B.

The study part B will be an efficacy and safety assessment of the dose of AVX-012 ophthalmic solution selected in the study part A (Low dose or High dose AVX-012) administered three times a day (TID) and twice a day (BID) when compared with the vehicle (placebo). Approximately 148 patients will be randomized 1:1:1:1 to study groups (Low dose or High dose AVX-012 and placebo [vehicle], TID and BID).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of at least 18 years of age.
* Diagnosis of dry eye (by a health care professional) for at least 3 months prior to screening visit.
* Normal lid anatomy.
* Intraocular pressure less than 22 mmHg (inclusive) in each eye.
* Best-corrected visual acuity measured by ETDRS in each eye of 20/200 (logMAR 1.0) or better.
* Schirmer I test score of ≥ 3 mm to ≤ 9 mm/ 5 min (with anesthesia).
* SANDE symptom score of 50 or more.
* Total ocular staining of minimum 1 in Oxford scale with fluorescein and/or green lissamine.
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.

Exclusion Criteria:

* History of other than dry eye, ocular surface of moderate to severe Meibomian gland disease (grades +++ to ++++ [moderately to severely altered expressibility and secretion quality]: moderate symptoms with mild to moderate corneal staining, mainly peripheral; or marked symptoms with marked corneal staining, central in addition), chronic, or acute ophthalmic disease in either eye, including glaucoma, macular degeneration, clinically significant cataract (primary or secondary).
* Best-corrected visual acuity score of 55 letters read or lower in each eye as measured by ETDRS (letters read method).
* Previous history of drug or any ingredient hypersensitivity.
* Intraocular or strabismus surgery or glaucoma laser surgery within the previous 6 months.
* History of refractive surgery in either eye (e.g., radial keratotomy, PRK, LASIK, etc.).
* Ocular trauma within the past 6 months.
* Relevant ocular pathology judged by the investigator such as; eyelid anomalies, corneal disorders, metaplasia of the ocular surface, current filamentous keratitis, or corneal neovascularization.
* Any history of herpes simplex or herpes zoster keratitis.
* Ocular infection (bacterial, viral, or fungal)
* Ocular medication of any kind, with the exception of artificial tears/gels/lubricants within the past 2 weeks of screening.
* Cyclosporine treatment during the 6 months prior to enrolment.
* Use of systemic medication that might cause dryness in the eye as a secondary effect (such as antihistaminics, hormone replacing therapies, etc.).
* Use of contact lens
* Use of additional artificial tears (other than study treatments) throughout the study, starting at screening visit.
* Participation in an investigational drug or device trial within the 30 days previous to screening visit.
* Any abnormality preventing reliable applanation tonometry of either eye.
* Central corneal thickness greater than 600 μm by conventional pachymetry.
* Signs of severe ocular surface diseases including corneal or conjunctival staining judged as severe by the investigator.
* Clinically significant systemic disease including uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular, endocrine disorders, previous cerebrovascular accident with a significant residual motor or sensory defect, progressive neurologic disorders (Parkinsonism, dementias, multiple sclerosis, unstable acquired seizure disorders) which might interfere with the study as judged by the investigator.
* Any systemic disease or medication that might course with known dryness in the eye.
* Changes of systemic medication that could have a substantial effect on intraocular pressure within 30 days prior to screening or anticipated during the study.
* Any medical condition (systemic or ophthalmic) that may, in the opinion of the investigator, preclude the safe administration of the investigational product or safe participation in this study.
* Pregnant or breastfeeding females or those with a positive pregnancy test.
* All females of childbearing potential must have a negative urine pregnancy test result at screening, and also agree to abstain from sexual intercourse with a male partner or agree to use a medically acceptable method of birth control (such as condom, diaphragm or cervical/vault cap with spermicide) until 28 days post-treatment. Males should also agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide until 28 days post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The objective of part A is to evaluate the safety of AVX-012 ophthalmic solution in subjects with dry eye syndrome. | 7 days (+1 day)
  Evaluation of vital signs (blood pressure and heart rate), laboratory analyses (haematology, biochemistry, and urine pregnancy test), best-corrected visual acuity (ETDRS), corneal anaesthesia (Cochet-Bonnet), intraocular pressure, biomicroscopy/staining (fluorescein), and ophthalmoscopy (dilated).
The objective of part B is to evaluate the efficacy of AVX-012 ophthalmic solution in treating symptoms of dry eye. | 28 days (+7 days)
  Percentage of patients achieving an improvement ≥ 20 points in the Symptom Assessment in Dry Eye (SANDE) questionnaire according to the different dosing frequencies (TID and BID).

SECONDARY OUTCOMES:
Confirm the safety of AVX-012 ophthalmic solution in subjects with dry eye syndrome. | 28 days (+7 days)
  Percentage of patients with adverse events from baseline (treatment period and post-treatment safety follow-up) according to the different dosing frequencies (TID and BID).
Change from baseline in corneal staining score | 28 days (+7 days)
Change from baseline in Schirmer I test score | 28 days (+7 days)
Change from baseline in tear film break up time score | 28 days (+7 days)
Change from baseline in conjunctival staining score | 28 days (+7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Tresserras, Study Director — Avizorex Pharma, S.L.
Locations (21):
- Spain (21):
  - Clinica Oftalvist Jerez, Jerez de la Frontera, Cadiz
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Clínica Oftalvist Vistahermosa, Alicante
  - Innova Ocular ICO Barcelona, Barcelona
  - Centro de Oftalmologia Barraquer, Barcelona
  - H Vall de Hebron, Barcelona
  - H Clinic, Barcelona
  - H General de Cataluña, Barcelona
  - H Germas Trias Pujol, Barcelona
  - clínica Oftalvist Granada, Granada
  - Clínica Universitaria de Navarra_ Madrid, Madrid
  - Clínica Oftalvist Moncloa, Madrid
  - H Universitario Ramón y Cajal, Madrid
  - H Clínico San Carlos, Madrid
  - Hospital General Universitario Reina Sofía, Murcia
  - Instituto Oftalmológico Fernández Vega, Oviedo
  - clinica Oftalvist Valencia, Valencia
  - Hospital Universitario La Fé, Valencia
  - Instituto Universitario de Oftalmobiología Aplicada (IOBA), Valladolid
  - H Miguel Servet, Zaragoza
  - H Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No